CLINICAL TRIAL: NCT03218345
Title: Multi-center Prospective Study on EUS-guided Radiofrequency Ablation for Solid Pancreatic Neoplasms
Brief Title: EUS-guided RFA for Pancreatic Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2015.531T
Record Dates: First submitted 2016-11-16; First posted 2017-07-14 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Neoplasms
Keywords: EUS-guided RFA; pancreatic ca; interventional EUS
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS-guided RFA (Experimental): EUS-guided RFA would be performed using a 19-gauge RFA electrode and a VIVA RF generator (STARmed, Korea)
  Interventions: Procedure: EUS-guided RFA

INTERVENTIONS:
Procedure: EUS-guided RFA — EUS-guided RFA would be performed using a 19-gauge RFA electrode and a generator

SUMMARY:
Radiofrequency ablation has been used for treatment of solid neoplasms of the liver, lung, kidney and adrenal. Recently, EUS-guided RFA has become available and the device allows EUS-guided treatment of pancreatic neoplasms. The procedure has been shown to be feasible in the porcine pancreas and was used to treat small groups of patients that are not suitable for surgery suffering from pancreatic neoplasms.

The aim of the current study is to perform a multi-center prospective study on EUS-guided radiofrequency ablation (RFA) of solid pancreatic neoplasms. The hypothesis is that EUS-guided RFA is safe, feasible and effective for treating solid pancreatic neoplasms.

DETAILED DESCRIPTION:
RFA causes tissue destruction through the application of a high frequency alternating current, generating local temperatures above 60°C and leading to coagulative necrosis. The technique has been widely used in many solid organ tumors and has been shown to result in 5-year survival rates comparable to surgery. The technique is currently the standard therapy in hepatocellular carcinoma and colorectal pulmonary metastasis particular in patients that are not suitable for surgery.

This study is a multi-center prospective study involving four high volume international institutions. Consecutive patients suffering from pancreatic neuroendocrine tumors and pancreatic cancers would be recruited. EUS-guided RFA would be performed using a 19-gauge RFA electrode and a generator. The primary outcome would be the overall adverse events rate. Secondary outcomes include mortality, technical success rate, completion ablation rate, 1 & 3 year overall and disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years-old or above
* Suffering from pancreatic neuroendocrine tumor or pancreatic ductal carcinoma (<5cm in largest diameter) that was confirmed by fine needle aspiration cytology
* Unsuitable for surgery, due to one (or more) of the following items:

  * ASA score > II*
  * An alternative advanced malignancy
  * Unsuitable for surgery upon expert's opinion for any other reason
* Healthy individuals who are not keen for surgical resection
* Eligible for endoscopic intervention
* Written informed consent

Exclusion Criteria:

* Coagulopathy (international normalized ratio >1.3, partial thromboplastin time greater than twice that of control), platelet count <50,000x103/uL
* Pregnancy
* Patients with a poor mental condition or mental retardation, unable to understand the nature and possible consequences of the study
* Patients unwilling to undergo follow-up assessments
* Patients with liver cirrhosis, portal hypertension and/or gastric varices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Severe adverse events | 30 days
  Adverse events specific to RFA would be graded according to the lexicon of endoscopic adverse events 24. Potential adverse events specific to RFA include: post-RFA syndrome, pancreatitis, pancreatic leak, thermal injury

SECONDARY OUTCOMES:
Technical success rates | 1 week
  defined as successful puncture of the lesion with the RFA needle and completion of the ablation cycle.
Procedural times | 1 day
  Duration of the procedure
Hospital stay | 30 days
  Duration of hospital stay
Radiological response | 1 year
  Based on modified RECIST criterion
Number of re-interventions | 1 year
  Number of re-interventions after the procedure
Survival | 3 years
  Duration of survival after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anthony YB Teoh, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided